CLINICAL TRIAL: NCT02388412
Title: Evaluating the Diagnostic Accuracy of 18F-sodium Fluoride Positron Emission Tomography for Identification of High-risk Vulnerable Coronary Atherosclerotic Plaque in Patients With Coronary Artery Disease
Brief Title: 18F-NaF-PET for Identification of TCFA
Acronym: NaF-PET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor of Internal Medicine and Cardiology Department, Seoul National University Hospital
Other Study IDs: NCT7895126
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Positron emission tomography; Tissue background ratio; Optical coherence tomography; Thin cap fibroous atheroma; Vulnerability; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Vulnerable plaque in optical coherence tomogrpahy: OCT-derived vulnerable plaque is defined as composite of thin-cap fibrous atheroma (cap thickness in optical coherence tomography < 60um), prominent macrophage, or prominent microvessels.
- Non-vulnerable plaque in Optical coherence tomogrpahy: OCT-derived vulnerable plaque is defined as composite of thin-cap fibrous atheroma (cap thickness in optical coherence tomography < 60um), prominent macrophage, or prominent microvessels. OCT-derived non-vulnerable plaque is defined as a plaque without any of the findings

SUMMARY:
Recently, positron emission tomography(PET) using 18F-Sodium fluoride (NaF) showed promising results for detecting vulnerable plaques in some pilot studies.

In this study, the investigators will evaluate the diagnostic accuracy of 18F-NaF PET for non-invasively detecting vulnerable plaque, diagnosed by optical coherence tomography (OCT).

DETAILED DESCRIPTION:
It has been well known that mechanism of acute coronary syndrome is plaque rupture and occlusion of coronary artery by this plaque rupture. Until now, evaluation of vulnerable plaque have been mainly performed with invasive imaging modalities such as optical coherence tomography or intravascular ultrasound.

Recently, positron emission tomography(PET) using 18F-Sodium fluoride (NaF) showed promising results for detecting vulnerable plaques in some pilot studies.

In this study, we will evaluate the diagnostic accuracy of 18F-NaF PET for non-invasively detecting vulnerable plaque, diagnosed by optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with angina pectoris who are scheduled to do invasive coronary angiography.
* 2. Patients who have moderate (40-70%) stenosis at proximal or mid-portion of major coronary arteries. Confirmed by coronary CT angiography.
* 3. Patients who are anticipated coronary artery disease.(Probability > 90 %)
* 4. Acute coronary syndrome.

Exclusion Criteria:

* 1. Stenosis at distal coronary or small vessel.
* 2. Patients who don't have moderate (40-70%) stenosis at proximal or mid-portion of major coronary arteries. Confirmed by invasive coronary angiography.
* 3. Inadequate quality of 18F-NaF PET-CT
* 4. Inadequate quality of Optical Coherence Tomography (OCT), IVUS, Coronary CT angiography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina pectoris
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Difference of tissue background ratio measured by 18F-NaF PET between Vulnerable and non-vulnerable plaque | up to 1 week
  Difference of tissue background ratio measured by 18F-NaF PET between Vulnerable and non-vulnerable plaque

SECONDARY OUTCOMES:
Differencce of Maximum SUV value between Vulnerable and non-vulnerable plaque | up to 1 week
  Tissue-to-background ratios were calculated for each participant by dividing the maximal SUV measured in aortic valves by the mean SUV of blood in inferior vena cava
Number of participants demonstrating at least 1 low-attenuation coronary atherosclerotic plaque | up to 1 week
  Number of participants demonstrating at least 1 low-attenuation coronary atherosclerotic plaque
Cardiac death and all-cause mortality | 1 year
  Between High-TBR and Low-TBR Plaque
Non-fatal target vessel myocardial infarction | 1 year
  Between High-TBR and Low-TBR Plaque
Target vessel revascularization | 1 year
  Between High-TBR and Low-TBR Plaque
Target vessel restenosis | 1 year
  Between High-TBR and Low-TBR Plaque

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Bon-Kwon, MD, PhD, Principal Investigator — Seoul National University Hospital; Paeng Jin Cheol, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JM, Bang JI, Koo BK, Hwang D, Park J, Zhang J, Yaliang T, Suh M, Paeng JC, Shiono Y, Kubo T, Akasaka T. Clinical Relevance of 18F-Sodium Fluoride Positron-Emission Tomography in Noninvasive Identification of High-Risk Plaque in Patients With Coronary Artery Disease. Circ Cardiovasc Imaging. 2017 Nov;10(11):e006704. doi: 10.1161/CIRCIMAGING.117.006704. PMID 29133478